CLINICAL TRIAL: NCT04747626
Title: B-SAFER: Branched Stented Anastomosis Frozen Elephant Trunk Repair
Acronym: B-SAFER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Roselli, M. D. (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor-Investigator, Eric Roselli, M. D., Sponsor/Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G200342
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Thoracic Aortic Aneurysm; Aortic Dissection; Congenital Aortic Anomaly
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Implantation of a physician-modified endovascular stentgraft(s) to treat the proximal aorta in subjects with aortic disease involving multiple segments.
  Interventions: Device: B-SAFER

INTERVENTIONS:
Device: B-SAFER — Simplified hybrid frozen elephant trunk repair will be performed by utilizing B-SAFER technique which involves a physician modified endovascular stentgraft to treat the proximal aorta in subjects with aortic disease involving multiple segments.

SUMMARY:
A prospective, single-center, non-blind, non-randomized safety and feasibility study of the hybrid repair of thoracic aortic pathologies requiring repair of the aortic arch proximal to the origin of innominate artery.

DETAILED DESCRIPTION:
The proposed Investigational Device Exemption (IDE) is to assess the safety and preliminary effectiveness of the simplified hybrid frozen elephant trunk repair technique Branched Stented Anastamosis Frozen Elephant Trunk Repair (B-SAFER) which involves a physician modified endovascular stentgraft to treat the proximal aorta in subjects with aortic disease involving multiple segments. The study will also evaluate the device functionality when using this operative technique for device implantation including multiple components.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Subject is willing and able to give written informed consent to participate in the study or the subject's legally authorized representative has given written informed consent for the subject to participate in the study.
3. Expected life expectancy of greater than two years after repair
4. Subject has aortic pathology and requires repair or replacement of multiple damaged or diseased segments of the thoracic aorta (at least one of the following condition): Thoracic aortic aneurysm considered at increased risk for rupture or complications, Acute aortic dissection requiring urgent repair, Congenital aortic disease requiring repair

Exclusion Criteria:

1. Subject is unfit for open surgical repair involving circulatory arrest
2. Subject is comatose or suffering from irreversible severe brain malperfusion
3. Subject has known sensitivity to components of the devices
4. Subject has an active systemic infection that, in the opinion of the investigator, would compromise the outcome of the surgical procedure
5. Subject is enrolled in another active study and has received an investigational product (device, pharmaceutical or biologic) within 6 months prior to the date of the implant or has not reached the primary endpoint of the study
6. Subject has an uncorrectable bleeding anomaly
7. Subject has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre- and post- procedure
8. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Up to 30 days
  Individual rate of occurrence of the death from all-cause
Stroke, excluding TIA | Up to 30 days
  Individual rate of occurrence of stroke
Paralysis, excluding paraparesis | Up to 30 days
  Individual rate of occurrence of paralysis
Technical success | 24 hours
  Composite of the following criteria: successful delivery of the device through the vasculature, successful deployment of the device at the intended location, and patient survival
Patency of all graft/endograft components | At hospital discharge or at 1 month
  Patent graft/endografts confirmed by CT imaging assessment
Complete sealing of the aortic pathology | At hospital discharge or 1 month
  Absence of Type Ia and IIIa/b endoleak, complete coverage of PAU cases, and isolation of the primary entry tear in dissection cases confirmed by CT imaging assessment

SECONDARY OUTCOMES:
Aortic related death | Up to 36 months after the index procedure
  Individual rate of the aortic related death
Pseudoaneurysm at the treatment sites | Up to 36 months after the index procedure
  Individual rate of the pseudoaneurysm at the treatment sites
Unanticipated aortic or branch-related re-operation | Up to 36 months after the index procedure
  Individual rate of the unanticipated aortic or branch-related re-operation
Late Type I endoleak | Up to 36 months after the index procedure
  Individual rate of the Type I endoleak confirmed by CT imaging assessment
Late Type III endoleak | Up to 36 months after the index procedure
  Individual rate of the Type III endoleak confirmed by CT imaging assessment
Non-cardiac/non-aortic re-operations | Up to 36 months after the index procedure
  Individual rate of non-cardiac/non-aortic re-operations
Vocal Cord paralysis | Up to 36 months after the index procedure
  Individual rate of vocal cord paralysis
Myocardial infarction | Up to 36 months after the index procedure
  Individual rate of myocardial infarction
Respiratory failure | Up to 36 months after the index procedure
  Individual rate of respiratory failure
Renal failure requiring dialysis | Up to 36 months after the index procedure
  Individual rate of renal failure requiring dialysis
Thromboembolic events | Up to 36 months after the index procedure
  Individual rate of thromboembolic events
Failed patencies in graft, or endovascular stent-graft including the branch(es) | Up to 36 months after the index procedure
  Individual rate of failed patencies in gaft or endovascular stent-graft including branch(es)
Secondary unplanned interventions in the treated vascular segment or related to the original pathology | Up to 36 months after the index procedure
  Individual rate of secondary unplanned interventions in the treated vascular segment or related to the original pathology
Aortic rupture | Up to 36 months after the index procedure
  Individual rate of aortic rupture
Device integrity failures | Up to 36 months after the index procedure
  Individual rate of device integrity failures confirmed by CT imaging assessment
Device crimping/kinking | Up to 36 months after the index procedure
  Individual rate of device crimping/kinking confirmed by CT imaging assessment
Device migration | Up to 36 months after the index procedure
  Individual rate of device migration (>10 mm based on the position of the device implantation) compared to baseline confirmed by CT imaging assessment
Thrombosis of the device lumen | Up to 36 months after the index procedure
  Individual rate of thrombosis of the device lumen confirmed by CT imaging assessment
Surgical graft/stentgraft infection | Up to 36 months after the index procedure
  Individual rate of surgical graft/stentgraft infection
Incidence of all endoleak types | Up to 36 months after the index procedure
  Individual rate of all endoleak types confirmed by CT imaging assessment
Migration of the distal extension | Up to 36 months after the index procedure
  Individual rate of distal extension migration (>10 mm based on the position of the device implantation) confirmed by CT imaging assessment
Non-serious and serious adverse events | Up to 36 months after the index procedure
  Individual rate of non-serious adverse events
Failure of device-extension integrity resulting in a compromised seal and blood leakage or movement of the device | Up to 36 months after the index procedure
  Individual rate of the extension device integrity issues confirmed by CT imaging assessment
Incidence of Type III endoleak related to the extension device | Up to 36 months after the index procedure
  Individual rate of the Type III endoleak related to the extension device confirmed by CT imaging assessment
Incidence of failed patency of the device-extension overlap | Up to 36 months after the index procedure
  Individual rate of failed patency of the device-extension overlap confirmed by CT imaging assessment
Incidence of MAE at 30 days post-extension | Up to 36 months after the index procedure
  Individual rate and type of MAE at 30 days post-extension
Incidence of secondary procedures related to the extension | Up to 36 months after the index procedure
  Individual rate secondary procedures related to the extension

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No